CLINICAL TRIAL: NCT05749640
Title: Clinical Evaluation of the Proximal Contact Tightness and Location in Class II Composite Restoration Using Different Contact Forming Instruments
Brief Title: The Proximal Contact Tightness and Location in Class II Composite Restorations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: karim mohamed (Other)
Responsible Party: Sponsor-Investigator, karim mohamed, Clinical instructor at faculty of dentistry Alexandria university, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AlexandriaU 0425-04/2022
Record Dates: First submitted 2022-10-24; First posted 2023-03-01 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Tooth Decay
MeSH Terms: conditions — Dental Caries | interventions — PERform Soft

STUDY DESIGN:
Intervention Model Description: This study will be a randomized control clinical trial in accordance with the Consolidated Standards of Reporting Trials (CONSORT) guidelines
Who Masked: Participant, Outcomes Assessor
Masking Description: Each case will be represented by a code and the group name. These will be sealed in a sequentially numbered opaque envelope and the set of envelopes will be given to the senior supervisor. When the investigator wants to enroll a new case, he will notify the supervisor who will take the next inline envelope and will write the name of the participant on it. At the time of intervention implementation, the investigator will open the sealed envelope and retrieve the allocation and apply.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Palodent® plus sectional matrix system "Control group" (Active Comparator)
  Interventions: Other: Precontoured sectional matrix EZ COAT
- PerForm™ "Experimental" (Experimental)
  Interventions: Other: PerForm™
- Trimax™ "Experimental" (Experimental)
  Interventions: Other: AdDent Trimax™
- Contact Pro™ "Experimental" (Experimental)
  Interventions: Other: Contact Pro™

INTERVENTIONS:
Other: Precontoured sectional matrix EZ COAT — All teeth will be treated with (Palodent ® plus sectional matrix system) (sectional matrix, biting ring, plastic diamond wedge)
  Arms: Palodent® plus sectional matrix system "Control group"
Other: PerForm™ — Treated with (PerForm™) as Contact Forming Instrument with (Palodent ® plus sectional matrix system)
  Arms: PerForm™ "Experimental"
Other: AdDent Trimax™ — Treated with (AdDent Trimax™) as Contact Forming Instrument with (Palodent ® plus sectional matrix system)
  Arms: Trimax™ "Experimental"
Other: Contact Pro™ — Treated with (Contact Pro™) as Contact Forming Instrument with (Palodent ® plus sectional matrix system)
  Arms: Contact Pro™ "Experimental"

SUMMARY:
This study aims to investigate consecutive biological changes in proximal contact tightness using digital force gauge and evaluate proximal contact location using cone beam computed tomography between class II direct composite restorations and adjacent teeth after using sectional matrix system and with different contact forming instruments.

ELIGIBILITY:
Inclusion Criteria:

* Presence of proximal caries in CBCT x-ray with score 3 to 4 according to the radiographic International Caries Detection and Assessment System (ICDAS).
* Presence of the antagonist and the adjacent tooth making contact.
* The teeth to be restored had to show no signs of pulpitis but positive sensitivity using endo ice testing.
* Size of the isthmus with no more than 2/3 of the intercuspal distance
* Good oral health and absence of periodontal disease
* Patients who are not suffering from severe systemic diseases or allergies

Exclusion Criteria:

* Medically compromised patients
* Clinical signs of bruxism, traumatic malocclusion
* Pregnant or breast feeding at the time of restoration placement
* Intolerance or allergy toward the applied restorative materials

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change in proximal contact tightness | baseline, immediately postoperative, 1 month, 3 month, 9 month, and 12 month
  Proximal contact tightness (PCT) will be measured using the custom-made contact pressure system that was based on the tooth pressure meter, a device fabricated at the University of Technology, Delft, the Netherlands. (20) The system will use a 0.05-mm-thick metal strip inserted interdentally from An occlusal direction . The metal strip will be connected to the digital force gauge (Mark-10 series 2 digital force gauge). The tightness of the proximal contact will be quantified as the maximum frictional force when the strip will slowly removed in a buccal-lingual direction. The maximum force will be recorded on the screen of the gauge for each measurement when the gauge will be switched to peak-mode

SECONDARY OUTCOMES:
Change in proximal contact location | baseline and immediately postoperative
  calibration will be carried out by a radiologist, who evaluates the teeth carefully scrolling down through the images from the floor of the pulp chamber in all three orthogonal reconstructions (axial, coronal, and sagittal). To ensure image standardization, all cone-beam computed tomography (CBCT) images will be chosen from a single machine with a standard field of view, voxel size, exposure time and the thickness of the slice.
  CBCT images will be analyzed with the built-in digital imaging software. The measurement tool will be used to determine the total length of the crown of the restored teeth, measured from the tip of the mesiobuccal cusp to the cementoenamel junction. Based on this length, the crown portion will be divided into three levels: coronal, middle and apical thirds.

CONTACTS AND LOCATIONS:
Locations (1):
- Karim Mohamed Wahba Abbass, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Abbassy KM, Elmahy WA, Holiel AA. Evaluation of the proximal contact tightness in class II resin composite restorations using different contact forming instruments: a 1-year randomized controlled clinical trial. BMC Oral Health. 2023 Oct 7;23(1):729. doi: 10.1186/s12903-023-03462-5. PMID 37805456